CLINICAL TRIAL: NCT02908958
Title: Clinical Study of Pegylated Somatropin (PEG Somatropin) to Treat Children Growth Hormone Deficiency: A Multicenter, Randomized, Parallel, Dose-control Clinical Trial II
Brief Title: Clinical Study of Pegylated Somatropin to Treat Children Growth Hormone Deficiency
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); The Second Hospital of Anhui Medical University (Other); Guangzhou Women and Children's Medical Center (Other); First People's Hospital of Hangzhou (Other); Qilu Hospital of Shandong University (Other); Zhejiang Provincial People's Hospital (Other); Zhejiang Provincial Hospital of TCM (Other); Central South University (Other); Southwest Hospital, China (Other); First Affiliated Hospital of Guangxi Medical University (Other); Shanghai Children's Medical Center (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); The First Affiliated Hospital of Xiamen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Xiangya Hospital of Central South University (Other); Shaoxing Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 004 CT-Zhejiang
Record Dates: First submitted 2016-09-19; First posted 2016-09-21 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2016-09

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEG-somatropin (Experimental): Low dose group, PEG Somatropin 0.14mg/kg/week, subcutaneous use, inject once a week, the duration is 26 weeks.
  Interventions: Biological: PEG-somatropin
- PEG-Somatropin (Experimental): High dose group, PEG Somatropin 0.2mg/kg/week, subcutaneous use, inject once a week, the duration is 26 weeks.
  Interventions: Biological: PEG-somatropin

INTERVENTIONS:
Biological: PEG-somatropin — High dose group: PEG Somatropin 0.2 mg/kg/w, subcutaneous use, inject once a week, the duration is for 26 weeks.
Biological: PEG-somatropin — Low dose group: PEG Somatropin 0.14 mg/kg/w, subcutaneous use, inject once a week, the duration is for 26 weeks.

SUMMARY:
To evaluate the safety and efficacy of PEG Somatropin Injection (Jintrolong®) in the treatment of short stature due to endogenous growth hormone deficiency (GHD) in the broad of population of children.

ELIGIBILITY:
Inclusion Criteria:

* Before starting treatment, the child is diagnosed as GHD according to medical history,clinical symptoms and signs, GH provocation tests and imaging examinators and other examinators.
* According to the height statistical data of Chinese children's physical development in nine cities in 2015, the height of the child is lower than the third percentile of normal children's growth curve in the same age and same gender.
* Height velocity (HV) ≤5.0 cm/yr.
* GH provocation tests with two different mechanisms showed that GH peak concentration of the child is < 10.0ng/ml.
* Bone age (BA) ≤9 years in girls or ≤ 10 years in boys, and the BA is 1 year less than the CA.
* Prepuberty status (Tanner I stage), age ≥3 years old, girls and boys are acceptable.
* The child did not receive the treatment of growth hormone within 6 months.
* Subjects are willing and able to cooperate to complete scheduled visits, treatment plans and laboratory tests and other procedures, and they sign informed consent.

Exclusion Criteria:

* The child is dysfunction of liver and kidney (ALT) 2 times of the upper limit of normal value, Cr> the upper limit of normal value).
* The child has positive hepatitis B core antibody (HBc), hepatitis B surface antigen (HBsAg) and hepatitis B e antigen (HBeAg).
* The child is known as hypersensitivity to PEG Somatropin.
* The child has severe cardiopulmonary, hematological diseases, malignant tumors, general infection or immunodeficiency diseases.
* The child has potential tumor (family history).
* The child has diabetics.
* The child has abnormal growth and development, such as Turner's syndrome, constitutional delay of growth and puberty, Laron syndrome, growth hormone receptor deficiency, short stature girls with potential chromosomal abnormalities.
* The child took part in other clinical trials within 3 months.
* Other conditions are excluded when the investigator preclude the enrollment into the study.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 900 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The change of Height Standard Deviation Score for Chronological Age before and after the treatment (ΔHtSDSCA) | 26 weeks
  HtSDSCA = (Height at the evaluated time point- the mean value of normal children in the same gender and same age) / the height SD of normal children in the same gender and same age

SECONDARY OUTCOMES:
HtSDSBA | 26 weeks
  HtSDSBA = (height at the evaluated time point-the mean value of normal children in the same gender and same age) / height SD of normal children in the same bone age and same gender
Annual height velocity | 26 weeks
  Annual Growth Velocity (cm/yr) = 12×(Height at the end of treatment-Height at the beginning of treatment)/the treatment duration (month)
Standard Deviation Score of serum IGF-1 (IGF-1 SDS) | 26 weeks
  IGF-1 SDS = (actual concentration of IGF-1-the median of IGF-1 concentration of normal children in the age and same gender) / SD of IGF-1 concentration of normal children in the same gender and same age
Bone Maturation | 26 weeks
  Bone Maturation = (BA at the end of treatment-BA at the beginning of treatment)/ the treatment duration (Year)

CONTACTS AND LOCATIONS:
Overall Officials: Junfen Fu, PhD, Principal Investigator — The Children's Hospital of Zhejiang University School of Medicine
Locations (22):
- China (22):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Wuhu No.1 People's Hospital, Wuhu, Anhui
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guangzhou Women and Children's Medical Center, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Harbin Children's Hospital, Harbin, Heilongjiang
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Children's Hospital of Changchun, Changchun, Jilin
  - Qilu Children's Hospital of Shandong University, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Chengdu Women and Children's Central Hospital, Chengdu, Sichuan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - The Children's Hospital ,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial Hospital of Traditional Chinese Medcine Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Ningbo Women and Children's Hospital, Ningbo, Zhejiang
  - Shaoxing Second Hospital, Shaoxing, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Southwest Hospital, Third Military Medical University, Chongqing
  - Shanghai Children's Medical Center, Shanghai

REFERENCES:
- [Derived] Jiang Z, Chen X, Dong G, Lou Y, Zhang J, Cheng X, Pan J, Liao W, Wu J, Huang X, Jin X, Liu D, Zeng T, Zhu S, Dong Q, Luo X, Lan D, Cao L, Zhang X, Liu J, Dai M, Zhang M, Liu L, Dong J, Zhao D, Ni S, Fu J. Short-term efficacy and safety of a lower dose of polyethylene glycol recombinant human growth hormone in children with growth hormone deficiency: A randomized, dose-comparison study. Front Pharmacol. 2022 Aug 11;13:955809. doi: 10.3389/fphar.2022.955809. eCollection 2022. PMID 36034802